CLINICAL TRIAL: NCT03744468
Title: Phase 1-2 Study Investigating Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of Various Combinations of BGB-A425 and LBL-007 With Tislelizumab in Patients With Advanced Solid Tumors
Brief Title: Study of BGB-A425 and LBL-007 in Combination With Tislelizumab in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-900-102; U1111-1278-0027 (Other: UTN Number); 2022-500694-14 (EudraCT Number)
Record Dates: First submitted 2018-10-17; First posted 2018-11-16 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Metastatic Solid Tumors for Phase 1,Dose Escalation and Phase 2 Safety Lead-in, HNSCC, NSCLC and RCC Participants for Phase 2
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicenter, nonrandomized Phase 1 and Phase 2 clinical trial. Phase 1 will determine the recommended phase 2 dose (RP2D) for the combination of BGB-A425 and Tislelizumab. Phase 2 safety lead-in will determine the RP2D for the combination of BGB-A425, Tislelizumab and/or LBL-007. Phase 2 dose expansion will continue to evaluate the safety but also focus on the efficacy of the double or triplet treatment combination in select tumor types.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Dose Escalation (Experimental): Dose escalation of BGB-A425 in combination with Tislelizumab in participants with advanced solid tumors
  Interventions: Drug: BGB-A425; Drug: Tislelizumab
- Phase 2 Safety Lead-in (Experimental): Dose escalation for Cohort A (LBL-007 + Tislelizumab) and Cohort B (BGB-A425 + LBL-007 + Tislelizumab) in participants with advanced solid tumors
  Interventions: Drug: BGB-A425; Drug: Tislelizumab; Drug: LBL-007
- Phase 2 Dose Expansion (Experimental): Further explore the safety and clinical activity of BGB-A425 and LBL-007 in combination with Tislelizumab in participants with NSCLC, HNSCC and RCC
  Interventions: Drug: BGB-A425; Drug: Tislelizumab; Drug: LBL-007

INTERVENTIONS:
Drug: BGB-A425 — Humanized IgG1-variant monoclonal antibody against TIM-3
  Other Names: Surzebiclimab
Drug: Tislelizumab — Humanized, IgG4-variant monoclonal antibody against PD-1
  Other Names: BGB-A317
Drug: LBL-007 — Human anti LAG-3 IgG4-kappa antibody
  Other Names: Alcestobart
  Arms: Phase 2 Dose Expansion; Phase 2 Safety Lead-in

SUMMARY:
This is an open-label, multicenter, nonrandomized Phase 1 and 2 clinical trial evaluating various combinations of BGB-A425 and/or LBL-007 with tislelizumab.

DETAILED DESCRIPTION:
Blocking antibodies targeting PD-1 have achieved remarkable results in the treatment of many types of tumors. However, based upon the rate of primary and secondary resistance to PD-1 blockade, it is apparent that additional immuno-regulatory mechanism(s) underlie tumor immune escape. Indeed, research shows that the TIM-3 pathway cooperates with PD-1 to maximize the suppression of effector TILs as well as promote resistance to anti-PD-1 therapy. Therefore, TIM-3 represents an ideal target with the potential to significantly improve and/or extend the therapeutic benefit of anti-PD-1 therapy to a greater number of patients.

TIM3, LAG3, and PD-1 function as immune checkpoint receptors in the overlapping regulation of immune tolerance and have been shown to be co-overexpressed on the tumor infiltrating lymphocytes (TILs) from the participant samples of various solid tumors. Furthermore, emerging clinical data and preclinical data demonstrate co-expression of Tim-3, LAG-3, PD-1 often yield T cells' exhausted immunophenotype (ie, cytokine expression, proliferation etc.). Cancer cells take advantage of PD-1, TIM-3, and LAG-3 in inhibiting immune cells' function, and escape the immune surveillance. Based upon the overlapping expression profiles and immuno-regulatory functions, TIM-3 and LAG-3 mediated adaptive resistance, there is strong scientific rationale that simultaneous targeting of these checkpoint blockers, could potentially increase therapeutic benefit and may help to overcome the resistance arising due to anti-PD-(L)-1 therapy. Hence, this study will evaluate the safety and preliminary efficacy of BGB-A425 (anti TIM-3), LBL-007 (Anti-LAG-3) in combination with tislelizumab (anti PD-1) in patients with advanced solid tumors

This is an open-label, multicenter, nonrandomized Phase 1 and Phase 2 clinical trial. Phase 1 will determine the recommended phase 2 dose (RP2D) for the combination of BGB-A425 and Tislelizumab. Phase 2 safety lead-in will determine the RP2D for the combination of BGB-A425, Tislelizumab and/or LBL-007. Phase 2 dose expansion will continue to evaluate the safety but also focus on the efficacy of the doublet or triplet treatment combination in select tumor types.

ELIGIBILITY:
Key Inclusion Criteria:

Has Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1.

* Adequate organ function
* Phase 1 Dose Escalation + Phase 2 Safety Lead-In: Participants with histologically or cytologically confirmed advanced, metastatic, unresectable solid tumors who have previously received standard systemic therapy or for which treatment is not available, not tolerated or refused.
* Phase 2 Dose-Expansion: Participants with one of the following histologically or cytologically confirmed solid tumors:
* For HNSCC participants in cohort 1,4 and 6 (PD-L1 positive):

Recurrent/metastatic head and neck squamous cell cancer of the oral cavity, oropharynx, hypopharynx, and/or larynx whose tumor is not amenable to local therapy with curative intent (ie, surgery or radiation therapy with or without chemotherapy • For NSCLC participants in Cohort 2, 5 and 7 (PD-L1 positive): Locally recurrent Stage IIIB, stage IIIC or Stage IV squamous or non-squamous non-small cell lung cancer

• For RCC participants in Cohort 3: Locally advanced unresectable or metastatic and histologically confirmed renal cell carcinoma with a clear cell histology

Key Exclusion Criteria:

* NSCLC patients with known EGFR mutation, BRAF mutation, ALK fusion, or ROS1 fusion
* Active leptomeningeal disease or uncontrolled, untreated brain metastasis.
* Active autoimmune diseases or history of autoimmune diseases that may relapse.
* Interstitial lung disease, noninfectious pneumonitis or uncontrolled lung diseases
* Uncontrolled diabetes or significant cardiac issues
* Infections requiring systemic antibacterial, antifungal, or antiviral therapy
* History of severe hypersensitivity reactions to other monoclonal antibodies
* History of HIV infection or untreated chronic hepatitis B or chronic hepatitis B virus carriers
* Major surgical procedure within 28 days before study drug administration
* Chemotherapy, radiotherapy, immunotherapy or any investigational therapies within 28 days (PH 2 Safety Lead-In) or 14 days (PH 2 Dose Expansion) or 5 half-lives of (whichever is shorter) of first administration of study drug(s).
* With infections (including tuberculosis infection, etc) requiring systemic antibacterial, antifungal, or antiviral therapy ≤ 14 days prior to the first dose of study drug(s), or a requirement for chronic prophylactic treatment with antibiotics.
* Concurrent participation in another therapeutic clinical trial
* Received prior therapies targeting TIM-3and/or LAG3

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Phase 1 Dose Escalation and Phase 2 Safety lead-in: Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Approximately 2 years
  A TEAE is defined as an AE that had an onset date or a worsening in severity from baseline (pretreatment) on or after the first dose of study drug up to 30 days following study drug discontinuation or initiation of new anticancer therapy, whichever comes first.
  An SAE is any untoward medical occurrence that at any dose results in death or is life threatening.
Phase 1 Dose Escalation: Maximum Tolerated Dose (MTD) | Approximately 2 years
  The MTD or MAD is defined as the highest dose at which < 33% of the participants experience a dose limiting toxicity (DLT)
Phase 2 Dose Expansion: Objective Response Rate (ORR) | Approximately 2 years
  ORR is determined from the investigator derived tumor assessments per RECIST v1.1

SECONDARY OUTCOMES:
Phase 1 and Phase 2 : Duration of Response (DOR) | Phase 1 or 2 Expansion - Approximately 2-3 years each
  Duration of response (DOR) will be determined from investigator derived tumor assessments per Response Evaluation Criteria in Solid Tumors (RECIST) v. 1.1.
Phase 1 and Phase 2 : Disease control rate (DCR) | Phase 1 or 2 Expansion - Approximately 2-3 years each
  Disease control rate (DCR) will be determined from investigator derived tumor assessments per Response Evaluation Criteria in Solid Tumors (RECIST) v. 1.1.
Phase 1 and Phase 2 : Progression free survival | Phase 2 Expansion - Approximately 3 years
  Progression free survival will be determined from investigator derived tumor assessments per RECIST 1.1.
Pharmacokinetic (PK) Parameter: Minimum Concentration (Cmin) of BGB-425 and LBL-007 | Phase 1 and Phase 2- Approximately 2-3 years each
PK Parameter: Area Under the Curve (AUC), 0 to 21 days of BGB-425 and LBL-007 | Phase 1 and Phase 2- Approximately 2-3 years each
PK Parameter: Maximum Concentration (Cmax) of BGB-425 and LBL-007 | Phase 1 and Phase 2- Approximately 2-3 years each
PK Parameter: Clearance (CL) of BGB-425 and LBL-007 | Phase 1 and Phase 2- Approximately 2-3 years each
PK Parameter: Volume of Distribution (Vz) of BGB-425 and LBL-007 | Phase 1 and Phase 2- Approximately 2-3 years each
PK Parameter: terminal half-life (t1/2) of BGB-425 and LBL-007 | Phase 1 and Phase 2- Approximately 2-3 years each
Percentage of participants with anti-BGB-A425 and LBL-007 antibodies | Phase 1 and Phase 2- Approximately 2-3 years each
Phase 2 Dose Expansion: Number of participants with TEAEs and SAEs including physical examinations, electrocardiograms and laboratory assessments | Phase 1 and Phase 2- Approximately 2-3 years each

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (42):
- United States (11):
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Weill Cornell Medical College Newyork Presbyterian Hospital, New York, New York
  - University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
  - Ut Health San Antonio Mays Cancer Center, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Schar Cancer Institute, Fairfax, Virginia
- Australia (11):
  - Sydney Southwest Private Hospital, Liverpool, New South Wales
  - Sunshine Coast Hospital and Health Service, Birtinya, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Calvary North Adelaide Hospital, North Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Cabrini Research and Education Institute, Malvern, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Western Health Sunshine Hospital, St Albans, Victoria
  - Hollywood Private Hospital, Nedlands, Western Australia
  - Linear Clinical Research, Nedlands, Western Australia
- France (2):
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Centre de Lutte Contre Le Cancer Francois Baclesse, Caen
- Italy (3):
  - Irccs Azienda Ospedaliero Universitaria Bologna, Bologna
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Istituto Di Candiolo Irccs, Torino
- Poland (2):
  - Centrum Onkologiiim Prof F Lukaszczyka Wbydgoszczy, Bydgoszcz
  - Narodowy Instytut Onkologii Im Marii Skodowskiej Curie Pastwowy Instytut Badawczy, Warsaw
- South Korea (8):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbukdo
  - The Catholic University of Korea, St Vincents Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Incheon Gwang'yeogsi
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, Seoul, Seoul Teugbyeolsi
  - Ulsan University Hospital, Donggu, Ulsan Gwang'yeogsi
- Spain (5):
  - Institut Catala Doncologia, Barcelona
  - Ico Hug Trias I Pujol, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Hm Madrid Sanchinarro, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/